CLINICAL TRIAL: NCT05541744
Title: The Use of Molecular Radiogenomics in Non-small Cell Lung Cancer
Acronym: NSCLC
Status: Recruiting | Type: Observational
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRB111-168-A
Record Dates: First submitted 2022-09-13; First posted 2022-09-15 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Lung Cancer
Keywords: non-small cell lung cancer; Radiogenomics; 18F-FDG PET; whole exome sequencing; molecular imaging
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Lung cancer is currently the leading cause of cancer-related mortality worldwide, and the dominant histopathology is non-small cell lung cancer (NSCLC). Although many new targeted and immunomodulation therapies have emerged, not all patients are responsive to novel therapeutics. A more reliable and accurate risk stratification model to predict the treatment response and survival outcomes are still lacking. The 18F-fluorodeoxyglucose (18F-FDG) positron emission tomography (PET) derived radiomics can be used to interrogate tumor biologies such as glycolytic activity and heterogeneity. It can, therefore, be used to predict treatment response and survival outcomes. Cancer genomics derived from gene sequencing can evaluate cancer's genetic alterations. It can be used to feature the genotype of the tumor. However, both tools have drawbacks; combining these two modalities may enable a more robust predictive model for more precise clinical decisions. During the investigator's former study project, the investigators published four Science Citation Index journal papers using the investigators' research results, which found that 18F-FDG PET radiomics can independently predict regional lymph node metastasis in NSCLC and cancer survival by stage. The preliminary findings of the investigator's former research project also disclosed an association between 18F-FDG PET-derived molecular radiomics with genomic heterogeneity and mutation of specific glucose metabolic genes. This time, the investigators plan to include deep radiomics in addition to traditional handcrafted radiomics. The investigators aim to investigate the radiogenomic patterns in different driver gene mutation statuses and clinical scenarios. Finally, the investigators seek to use radiogenomics as a prognostic stratification tool in patients with NSCLC.

DETAILED DESCRIPTION:
This is a prospective study and The investigators use routine pathological specimens for whole exome sequencing (WES) and immunohistochemical stains.

Pathological examinations include PD-L1, EGFR status, ALK, and ROS-1.

WES： Total DNA were extracted from paraffin-embedded tumor specimens with the QIAamp DNA FFPE Tissue Kit (QIAGEN GmbH, Hilden, Germany). The coding size was 45 Mb. For DNA whole exome sequence, briefly, tumors were sonicated by Covaris M220 sonicator (Life Technologies Europe, Gent, Belgium) and then ligated to adaptor for further amplification (Illumina® TruSeq Exome Library Prep, USA). After library preparation, all samples were sequenced using the NextSeq500 system according to the manufacturer's instructions (Illumina, San Diego, USA). The investigators run sequencing with 12 samples simultaneously (a total of 100 Gb). The sequence length was 150 bp with a paired-end (2*150bp). The average depth of sequencing is 100X. After sequencing performance, quality of reads file (fastq) was assessed by FastQC and then mapped using human Hg19 as the reference. Bam files were used as input for the Varscan algorithm to identify germline and somatic mutations. Variants annotated and filtered are manually checked using IGV (Integrative Genomics Viewer), then confirmed by Sanger sequence. The investigators analyze the clinical related gene alterations including actionable gene mutations (EGFR, BRAF, KRAS, and MET.) Also, clinically important genes including the mutation status of TP53 and SDH genes are analyzed. The investigators also analyzed the mutation status of glucose metabolic cluster genes.

TMB (tumor mutation burden) per megabase: The total number of mutations counted is divided by the size of the coding region of the targeted territory.

MATH (mutant-allele tumor heterogeneity): The investigators first obtain the MAF (the fraction of DNA that shows the mutated allele at a gene locus) of each tumor specimen. The MAF distribution will be used to calculate the median (center of distribution) and the MD (median deviation) of MAFs in a tumor. The MD is determined by obtaining the absolute differences of all MAFs from the median MAF. Then the median of the absolute differences is multiplied by a factor of 1.4826 to obtain the MD. The MATH is calculated as the percentage ratio of the MD to the median: MATH = (MD/median)×100 [45].

Shannon diversity index (Shannon entropy) [50]: The MAF distribution (histogram) of each patient's tumor specimen was obtained with different bin sizes (total bin size = S). The Shannon diversity index is then calculated according to the distribution of probabilities of each MAF bin.

The image features of FDG PET the investigators extracted as follows, <Handcrafted radiomics> The traditional image parameters include SUVmax, metabolic tumor volume (MTV) and total lesion glycolysis (TLG) of the primary tumor. The traditional FDG PET parameters are calculated using commercialized software (PBAS, PMOD 4.0). Radiomics (texture analysis) will be calculated only for pre-treatment FDG PET. The matrices of radiomic analysis include histogram analysis, Gray-level co-occurrence matrix (GLCM), gray-level run-length matrix (GLRLM), gray-level size zone matrix (GLSZM), neighborhood gray-tone difference matrix (NGTDM), and shape features.

<Deep radiomics> The investigators put the segmented volume into convolutional neural network (CNN) for analysis. The investigators will use supervised CNN to analyze the relationship between imaging with other outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 20-years
* Pathological proven non-small cell lung cancer and received complete staging work-up
* Pre-treatment pathological specimen of the primary tumor

Exclusion Criteria:

* Coexistence of non-aerodigestive tract cancer.
* Unable to comply to FDG PET/CT exam or poor image quality
* Unable to determine the primary tumor

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-small cell lung cancer, and able to be analyzed with radiomics of FDG PET and primary tumor whole exome sequencing.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Prognosis | three years
  Study the association of radiogenomics with the treatment response and survival

SECONDARY OUTCOMES:
Correlation of radiogenomics | one year
  Study the correlation of radiomics and genomics and pathological features

CONTACTS AND LOCATIONS:
Locations (1):
- Hualien Tzu Chi Hospital, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: No